CLINICAL TRIAL: NCT01805856
Title: Antimicrobial Prophylaxis for the Prevention of Surgical Site Infection in Thyroid and Parathyroid Surgery
Brief Title: Antimicrobial Prophylaxis in Thyroid and Parathyroid Surgery
Acronym: Ito-RCT1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ito Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ito-RCT1
Record Dates: First submitted 2013-03-05; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Thyroid Disease; Parathyroid Disease
Keywords: antimicrobial prophylaxis; AMP; surgical site infection; SSI; thyroid; thyroidectomy; parathyroid; surgery
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Diseases; Surgical Wound Infection | interventions — Piperacillin; Cefazolin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (intervention PIPC) (Experimental): Patients in group A (intervention PIPC) were given AMP of 2g PIPC intravenously just after intubation. If the operation time was longer than 3 hours, additional infusion of same dose PIPC was done. After coming back to the patients' own room, one more infusion of same dose of same drug was done.
  Interventions: Drug: PIPC piperacillin sodium
- Group B (intervention CEZ) (Experimental): Patients in Group B (intervention CEZ) were given AMP of 1g CEZ intravenously just after intubation. If the operation time was longer than 3 hours, additional infusion of same dose CEZ was done. After coming back to the patients' own room, one more infusion of same dose of same drug was done.
  Interventions: Drug: CEZ, cefazolin sodium
- Group C (without AMP) (No Intervention): Patients in Group C underwent surgery without any AMP.

INTERVENTIONS:
Drug: PIPC piperacillin sodium
  Other Names: PIPC, piperacillin sodium
  Arms: Group A (intervention PIPC)
Drug: CEZ, cefazolin sodium
  Arms: Group B (intervention CEZ)

SUMMARY:
The effectiveness of antimicrobial prophylaxis (AMP) for prevention of surgical site infection (SSI) following thyroid and parathyroid surgery remains uncertain. Present prospective randomized control study (Ito-RCT1) assessed the effectiveness of AMP in clean neck surgery associated with thyroid and parathyroid disease.

DETAILED DESCRIPTION:
Between November 2010 and April 2012, 2164 consecutive patients who agreed to attend the randomized control study were enrolled. All the participants received surgery for thyroid and parathyroid disease at Ito Hospital and randomized in three groups; Group A (n=541): operation with AMP (PIPC, piperacillin sodium), Group B (n=541): operation with AMP (CEZ, cefazolin sodium), and Group C (n=1082): operation without AMP.

Exclusion criteria

* Patients who did not agree to attend the randomized control study.
* Patients who received the operation including mediastinum with sternotomy.
* Patients who received the operation including additional resection of trachea, esophagus and larynx.
* Patients who received the re-operation for post-operative bleedings.
* Patients who had known allergy to cephem or penicillin.

ELIGIBILITY:
Inclusion Criteria:

* Between November 2010 and April 2012, 2164 consecutive patients who agreed to attend the randomized control study were enrolled. All the participants received surgery for thyroid and parathyroid disease at Ito Hospital.

Exclusion Criteria:

* Patients who did not agree to attend the randomized control study.
* Patients who received the operation including mediastinum with sternotomy.
* Patients who received the operation including additional resection of trachea, esophagus and larynx.
* Patients who received the re-operation for post-operative bleedings.
* Patients who had known allergy to cephem or penicillin.

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2164 (Actual)
Dates: Start 2010-11; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Surgical site infections after thyroid and parathyroid surgery | 1 month after operation
  Surgical site infection was defined as patients who are necessary to receive the treatment such as surgical drainage or antibiotic medication. When the patients receive the surgical drainage, microbial culture was performed.

SECONDARY OUTCOMES:
Side effect of the drug for Antimicrobial prophylaxis | 4 days after operation
  The appearances of drug allergic reactions (skin rash and anaphylactic shock) were checked at operating room. Blood test to check up liver and renal dysfunction was done on the 3rd POD. Liver and renal dysfunction is clinically diagnosed by patients' own physicians and the author, and only counted the cases which function got worse compared to preoperative data.

OTHER OUTCOMES:
Urinary tract infection after operation with or without antimicrobial prophylaxis | 1month after operation
  If the patients had a symptom of urinary tract infection, additional blood test and urine test were done to diagnose infection accurately.

CONTACTS AND LOCATIONS:
Overall Officials: Takashi Uruno, MD, Principal Investigator — Ito Hospital
Locations (1):
- Ito Hospital, Tokyo, Japan